CLINICAL TRIAL: NCT06491732
Title: Electrical Impedance Myography Via the Myolex mScan as an ALS Biomarker
Brief Title: EIM Via the Myolex mScan as an ALS Biomarker
Acronym: ElectricALS
Status: Recruiting | Type: Observational
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Seward Rutkove, Principal Investigator, Beth Israel Deaconess Medical Center
Other Study IDs: 2024P000292; HT9425-24-1-0650 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2024-07-01; First posted 2024-07-09 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Amyotrophic Lateral Sclerosis; Electrical Impedance Myography; Biomarker
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Amyotrophic Lateral Sclerosis: Patients diagnosed with ALS
  Interventions: Device: Electrical Impedance Myography

INTERVENTIONS:
Device: Electrical Impedance Myography — EIM is an impedance-based technology in which an imperceptible, high-, multi-frequency (e.g., 1 kHz to 10 MHz) electrical current is applied across two electrodes; the resulting voltage signals are measured across two sense electrodes
  Other Names: Myolex mScan

SUMMARY:
Amyotrophic lateral sclerosis (ALS) has been traditionally considered incurable and untreatable. But starting in the 1990s with the introduction of Riluzole, therapies are being discovered and ultimately approved for slowing disease progression. Many pharmaceutical companies continue to seek new therapeutic approaches. One critical aspect of all clinical trials is the need track to progression sensitively to identify the impact of therapy. Tools to track ALS progression must be convenient, objective, require minimal training, be easily standardized, cost-efficient, and have the potential to be applied effectively at home. There has been a push to identify accurate, objective biomarkers of ALS progression. In this study, the investigators propose to use Electrical impedance myography (EIM) to evaluate the progression of the disease. Work has shown that the EIM 50 kilohertz (kHz) phase value from one or more muscles, followed sequentially, can serve as an effective overall biomarker for assessing the rate of ALS progression for a single person.

DETAILED DESCRIPTION:
Amyotrophic lateral sclerosis (ALS) has been traditionally considered incurable and untreatable. But starting in the 1990s with the introduction of Riluzole, therapies are being discovered and ultimately approved for slowing disease progression. Given ALS's uniquely devastating nature, the fact that it is considered an "orphan disease", and uncertainties about its complex pathogenesis, many pharmaceutical companies continue to seek new therapeutic approaches. In fact, despite a relatively poor track record of success, there are a plethora of new studies starting up or planned in the near future. One critical aspect of all clinical trials is the need track to progression sensitively to identify the impact of therapy. Tools to track ALS progression must be convenient, objective (i.e. not influenced by patient or evaluator mood or engagement), require minimal training, be easily standardized, and be cost-efficient. Moreover, ideally, such measures, also called biomarkers, could also be used flexibly for improving individual patient care and could be applied effectively at home. Most ALS studies over the past two decades have relied on the ALS functional rating scale-revised (ALSFRS-R). Yet, it is relatively insensitive to change, altering, on average, less than 1 point per month, and requiring a large sample size to detect a drug effect, as demonstrated by several recent trials that have used it. There has been a push to identify accurate, objective biomarkers of ALS progression. In this study, the investigators propose to use Electrical impedance myography (EIM) to evaluate the progression of the disease. Work has shown that the EIM 50 kHz phase value from one or more muscles, followed sequentially, can serve as an effective overall biomarker for assessing the rate of ALS progression for a single person.

Aim 1: To evaluate the sensitivity of EIM 50 kHz phase values to ALS progression, as measured by the Myolex mScan device, such that it may be able to serve as a monitoring, prognostic, or pharmacodynamic biomarker in future studies of ALS.

Aim 2: To evaluate the potential for additional at-home assessments to improve sensitivity to change/deterioration in ALS and to assess general acceptability to patients/caregivers of doing these measurements at home.

Aim 3: To utilize the full set of multifrequency parameters to assess disease progression overtime via the application of machine learning analytics to increase the power of EIM as an ALS biomarker.

ELIGIBILITY:
Inclusion Criteria:

* Sporadic or familial ALS diagnosed as clinically possible, probable, lab-supported probable, or deﬁnite ALS deﬁned by revised El Escorial criteria
* Capable of providing informed consent and complying with study procedures in the investigator's opinion
* Time since ALS symptom onset ≤36 months
* Vital Capacity of ≥50% of predicted capacity as measured by forced vital capacity
* Must have a study partner for home visits
* Access to the internet for data upload
* Age 18 years or older

Exclusion Criteria:

* Clinically signiﬁcant unstable medical condition (other than ALS) that would affect the participant's ability to participate, according to the investigator's judgment
* Patient with pure upper motor neuron disease (PLS)
* Known history of unstable psychiatric disease, cognitive impairment, dementia, or active substance abuse
* Significant pitting edema (2+ or more) that would interfere with EIM measures
* Active cancer or history of cancer treated with chemotherapy and/or radiation
* BMI >35

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with ALS
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
EIM phase change over time | 8 months
  Mean and standard deviation in rate of change in EIM phase values compared to mean and standard deviation in rate of change in ALSFRS-R over 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Seward Rutkove, MD, Principal Investigator — Beth Israel Deaconess Medical Center; Masumeh Hatami, MD, Study Director — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
All de-identified data will be shared publicly through existing websites (such as the Pooled Resource Open-Access ALS Clinical Trials database). We will include relevant clinical and demographic information (all de-identified). The Digital Object Identifier (DOI) will be referenced in any publication to allow the research community easy access to the exact data used in the publication. The results of the study will also be shared via publication in open-access journals and at national and international ALS meetings (e.g., at the international ALS Motor Neuron Diseases meeting).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Upon completion and primary analysis of the study
Access Criteria: Public

REFERENCES:
- [Background] Bowser R, Cudkowicz M, Kaddurah-Daouk R. Biomarkers for amyotrophic lateral sclerosis. Expert Rev Mol Diagn. 2006 May;6(3):387-98. doi: 10.1586/14737159.6.3.387. PMID 16706741
- [Background] Mancuso R, Navarro X. Amyotrophic lateral sclerosis: Current perspectives from basic research to the clinic. Prog Neurobiol. 2015 Oct;133:1-26. doi: 10.1016/j.pneurobio.2015.07.004. Epub 2015 Aug 5. PMID 26253783
- [Background] Malik R, Lui A, Lomen-Hoerth C. Amyotrophic lateral sclerosis. Semin Neurol. 2014 Nov;34(5):534-41. doi: 10.1055/s-0034-1396007. Epub 2014 Dec 17. PMID 25520025
- [Background] DeJesus-Hernandez M, Mackenzie IR, Boeve BF, Boxer AL, Baker M, Rutherford NJ, Nicholson AM, Finch NA, Flynn H, Adamson J, Kouri N, Wojtas A, Sengdy P, Hsiung GY, Karydas A, Seeley WW, Josephs KA, Coppola G, Geschwind DH, Wszolek ZK, Feldman H, Knopman DS, Petersen RC, Miller BL, Dickson DW, Boylan KB, Graff-Radford NR, Rademakers R. Expanded GGGGCC hexanucleotide repeat in noncoding region of C9ORF72 causes chromosome 9p-linked FTD and ALS. Neuron. 2011 Oct 20;72(2):245-56. doi: 10.1016/j.neuron.2011.09.011. Epub 2011 Sep 21. PMID 21944778
- [Background] Renton AE, Majounie E, Waite A, Simon-Sanchez J, Rollinson S, Gibbs JR, Schymick JC, Laaksovirta H, van Swieten JC, Myllykangas L, Kalimo H, Paetau A, Abramzon Y, Remes AM, Kaganovich A, Scholz SW, Duckworth J, Ding J, Harmer DW, Hernandez DG, Johnson JO, Mok K, Ryten M, Trabzuni D, Guerreiro RJ, Orrell RW, Neal J, Murray A, Pearson J, Jansen IE, Sondervan D, Seelaar H, Blake D, Young K, Halliwell N, Callister JB, Toulson G, Richardson A, Gerhard A, Snowden J, Mann D, Neary D, Nalls MA, Peuralinna T, Jansson L, Isoviita VM, Kaivorinne AL, Holtta-Vuori M, Ikonen E, Sulkava R, Benatar M, Wuu J, Chio A, Restagno G, Borghero G, Sabatelli M; ITALSGEN Consortium; Heckerman D, Rogaeva E, Zinman L, Rothstein JD, Sendtner M, Drepper C, Eichler EE, Alkan C, Abdullaev Z, Pack SD, Dutra A, Pak E, Hardy J, Singleton A, Williams NM, Heutink P, Pickering-Brown S, Morris HR, Tienari PJ, Traynor BJ. A hexanucleotide repeat expansion in C9ORF72 is the cause of chromosome 9p21-linked ALS-FTD. Neuron. 2011 Oct 20;72(2):257-68. doi: 10.1016/j.neuron.2011.09.010. Epub 2011 Sep 21. PMID 21944779
- [Background] Gurney ME, Pu H, Chiu AY, Dal Canto MC, Polchow CY, Alexander DD, Caliendo J, Hentati A, Kwon YW, Deng HX, et al. Motor neuron degeneration in mice that express a human Cu,Zn superoxide dismutase mutation. Science. 1994 Jun 17;264(5166):1772-5. doi: 10.1126/science.8209258.
- [Background] Woolley SC, Strong MJ. Frontotemporal Dysfunction and Dementia in Amyotrophic Lateral Sclerosis. Neurol Clin. 2015 Nov;33(4):787-805. doi: 10.1016/j.ncl.2015.07.011. Epub 2015 Sep 8. PMID 26515622
- [Background] Walhout R, Verstraete E, van den Heuvel MP, Veldink JH, van den Berg LH. Patterns of symptom development in patients with motor neuron disease. Amyotroph Lateral Scler Frontotemporal Degener. 2018 Feb;19(1-2):21-28. doi: 10.1080/21678421.2017.1386688. Epub 2017 Oct 16. PMID 29037065
- [Background] Writing Group; Edaravone (MCI-186) ALS 19 Study Group. Safety and efficacy of edaravone in well defined patients with amyotrophic lateral sclerosis: a randomised, double-blind, placebo-controlled trial. Lancet Neurol. 2017 Jul;16(7):505-512. doi: 10.1016/S1474-4422(17)30115-1. Epub 2017 May 15. PMID 28522181
- [Background] Paganoni S, Macklin EA, Hendrix S, Berry JD, Elliott MA, Maiser S, Karam C, Caress JB, Owegi MA, Quick A, Wymer J, Goutman SA, Heitzman D, Heiman-Patterson T, Jackson CE, Quinn C, Rothstein JD, Kasarskis EJ, Katz J, Jenkins L, Ladha S, Miller TM, Scelsa SN, Vu TH, Fournier CN, Glass JD, Johnson KM, Swenson A, Goyal NA, Pattee GL, Andres PL, Babu S, Chase M, Dagostino D, Dickson SP, Ellison N, Hall M, Hendrix K, Kittle G, McGovern M, Ostrow J, Pothier L, Randall R, Shefner JM, Sherman AV, Tustison E, Vigneswaran P, Walker J, Yu H, Chan J, Wittes J, Cohen J, Klee J, Leslie K, Tanzi RE, Gilbert W, Yeramian PD, Schoenfeld D, Cudkowicz ME. Trial of Sodium Phenylbutyrate-Taurursodiol for Amyotrophic Lateral Sclerosis. N Engl J Med. 2020 Sep 3;383(10):919-930. doi: 10.1056/NEJMoa1916945. PMID 32877582
- [Background] Nikitin D, Makam AN, Suh K, McKenna A, Carlson JJ, Richardson M, Rind DM, Pearson SD. The effectiveness and value of AMX0035 and oral edaravone for amyotrophic lateral sclerosis: A summary from the Institute for Clinical and Economic Review's Midwest Comparative Effectiveness Public Advisory Council. J Manag Care Spec Pharm. 2023 Feb;29(2):216-221. doi: 10.18553/jmcp.2023.29.2.216. PMID 36705279
- [Background] Miller TM, Cudkowicz ME, Genge A, Shaw PJ, Sobue G, Bucelli RC, Chio A, Van Damme P, Ludolph AC, Glass JD, Andrews JA, Babu S, Benatar M, McDermott CJ, Cochrane T, Chary S, Chew S, Zhu H, Wu F, Nestorov I, Graham D, Sun P, McNeill M, Fanning L, Ferguson TA, Fradette S; VALOR and OLE Working Group. Trial of Antisense Oligonucleotide Tofersen for SOD1 ALS. N Engl J Med. 2022 Sep 22;387(12):1099-1110. doi: 10.1056/NEJMoa2204705. PMID 36129998
- [Background] Kiernan MC, Vucic S, Talbot K, McDermott CJ, Hardiman O, Shefner JM, Al-Chalabi A, Huynh W, Cudkowicz M, Talman P, Van den Berg LH, Dharmadasa T, Wicks P, Reilly C, Turner MR. Improving clinical trial outcomes in amyotrophic lateral sclerosis. Nat Rev Neurol. 2021 Feb;17(2):104-118. doi: 10.1038/s41582-020-00434-z. Epub 2020 Dec 18. PMID 33340024
- [Background] Ashhurst JF, Tu S, Timmins HC, Kiernan MC. Progress, development, and challenges in amyotrophic lateral sclerosis clinical trials. Expert Rev Neurother. 2022 Nov-Dec;22(11-12):905-913. doi: 10.1080/14737175.2022.2161893. Epub 2023 Jan 18. PMID 36543326
- [Background] Martinez-Gonzalez L, Martinez A. Emerging clinical investigational drugs for the treatment of amyotrophic lateral sclerosis. Expert Opin Investig Drugs. 2023 Feb;32(2):141-160. doi: 10.1080/13543784.2023.2178416. Epub 2023 Feb 16. PMID 36762798
- [Background] Paganoni S, Berry JD, Quintana M, Macklin E, Saville BR, Detry MA, Chase M, Sherman AV, Yu H, Drake K, Andrews J, Shefner J, Chibnik LB, Vestrucci M, Cudkowicz ME; Healey ALS Platform Trial Study Group. Adaptive Platform Trials to Transform Amyotrophic Lateral Sclerosis Therapy Development. Ann Neurol. 2022 Feb;91(2):165-175. doi: 10.1002/ana.26285. Epub 2022 Jan 10. PMID 34935174
- [Background] Cedarbaum JM, Stambler N, Malta E, Fuller C, Hilt D, Thurmond B, Nakanishi A. The ALSFRS-R: a revised ALS functional rating scale that incorporates assessments of respiratory function. BDNF ALS Study Group (Phase III). J Neurol Sci. 1999 Oct 31;169(1-2):13-21. doi: 10.1016/s0022-510x(99)00210-5. PMID 10540002
- [Background] Cudkowicz ME, Titus S, Kearney M, Yu H, Sherman A, Schoenfeld D, Hayden D, Shui A, Brooks B, Conwit R, Felsenstein D, Greenblatt DJ, Keroack M, Kissel JT, Miller R, Rosenfeld J, Rothstein JD, Simpson E, Tolkoff-Rubin N, Zinman L, Shefner JM; Ceftriaxone Study Investigators. Safety and efficacy of ceftriaxone for amyotrophic lateral sclerosis: a multi-stage, randomised, double-blind, placebo-controlled trial. Lancet Neurol. 2014 Nov;13(11):1083-1091. doi: 10.1016/S1474-4422(14)70222-4. Epub 2014 Oct 5. PMID 25297012
- [Background] Shefner JM, Wolff AA, Meng L, Bian A, Lee J, Barragan D, Andrews JA; BENEFIT-ALS Study Group. A randomized, placebo-controlled, double-blind phase IIb trial evaluating the safety and efficacy of tirasemtiv in patients with amyotrophic lateral sclerosis. Amyotroph Lateral Scler Frontotemporal Degener. 2016 Jul-Aug;17(5-6):426-435. doi: 10.3109/21678421.2016.1148169. Epub 2016 Mar 16. PMID 26982815
- [Background] Fournier CN, Bedlack R, Quinn C, Russell J, Beckwith D, Kaminski KH, Tyor W, Hertzberg V, James V, Polak M, Glass JD. Development and Validation of the Rasch-Built Overall Amyotrophic Lateral Sclerosis Disability Scale (ROADS). JAMA Neurol. 2020 Apr 1;77(4):480-488. doi: 10.1001/jamaneurol.2019.4490. PMID 31886839
- [Background] Visser J, Mans E, de Visser M, van den Berg-Vos RM, Franssen H, de Jong JM, van den Berg LH, Wokke JH, de Haan RJ. Comparison of maximal voluntary isometric contraction and hand-held dynamometry in measuring muscle strength of patients with progressive lower motor neuron syndrome. Neuromuscul Disord. 2003 Nov;13(9):744-50. doi: 10.1016/s0960-8966(03)00135-4. PMID 14561498
- [Background] Andres PL, Skerry LM, Munsat TL, Thornell BJ, Szymonifka J, Schoenfeld DA, Cudkowicz ME. Validation of a new strength measurement device for amyotrophic lateral sclerosis clinical trials. Muscle Nerve. 2012 Jan;45(1):81-5. doi: 10.1002/mus.22253. PMID 22190312
- [Background] Vender RL, Mauger D, Walsh S, Alam S, Simmons Z. Respiratory systems abnormalities and clinical milestones for patients with amyotrophic lateral sclerosis with emphasis upon survival. Amyotroph Lateral Scler. 2007 Feb;8(1):36-41. doi: 10.1080/17482960600863951. PMID 17364434
- [Background] Turner MR, Kiernan MC, Leigh PN, Talbot K. Biomarkers in amyotrophic lateral sclerosis. Lancet Neurol. 2009 Jan;8(1):94-109. doi: 10.1016/S1474-4422(08)70293-X. PMID 19081518
- [Background] Lu CH, Macdonald-Wallis C, Gray E, Pearce N, Petzold A, Norgren N, Giovannoni G, Fratta P, Sidle K, Fish M, Orrell R, Howard R, Talbot K, Greensmith L, Kuhle J, Turner MR, Malaspina A. Neurofilament light chain: A prognostic biomarker in amyotrophic lateral sclerosis. Neurology. 2015 Jun 2;84(22):2247-57. doi: 10.1212/WNL.0000000000001642. Epub 2015 May 1. PMID 25934855
- [Background] Shepheard SR, Wuu J, Cardoso M, Wiklendt L, Dinning PG, Chataway T, Schultz D, Benatar M, Rogers ML. Urinary p75ECD: A prognostic, disease progression, and pharmacodynamic biomarker in ALS. Neurology. 2017 Mar 21;88(12):1137-1143. doi: 10.1212/WNL.0000000000003741. Epub 2017 Feb 22. PMID 28228570
- [Background] Grolez G, Moreau C, Danel-Brunaud V, Delmaire C, Lopes R, Pradat PF, El Mendili MM, Defebvre L, Devos D. The value of magnetic resonance imaging as a biomarker for amyotrophic lateral sclerosis: a systematic review. BMC Neurol. 2016 Aug 27;16(1):155. doi: 10.1186/s12883-016-0672-6. PMID 27567641
- [Background] Alshikho MJ, Zurcher NR, Loggia ML, Cernasov P, Chonde DB, Izquierdo Garcia D, Yasek JE, Akeju O, Catana C, Rosen BR, Cudkowicz ME, Hooker JM, Atassi N. Glial activation colocalizes with structural abnormalities in amyotrophic lateral sclerosis. Neurology. 2016 Dec 13;87(24):2554-2561. doi: 10.1212/WNL.0000000000003427. Epub 2016 Nov 11. PMID 27837005
- [Background] Brown WF. A method for estimating the number of motor units in thenar muscles and the changes in motor unit count with ageing. J Neurol Neurosurg Psychiatry. 1972 Dec;35(6):845-52. doi: 10.1136/jnnp.35.6.845. PMID 4647858
- [Background] Shefner JM. Motor unit number estimation in human neurological diseases and animal models. Clin Neurophysiol. 2001 Jun;112(6):955-64. doi: 10.1016/s1388-2457(01)00520-x. PMID 11377252
- [Background] Swash M, de Carvalho M. The Neurophysiological Index in ALS. Amyotroph Lateral Scler Other Motor Neuron Disord. 2004 Sep;5 Suppl 1:108-10. doi: 10.1080/17434470410020067. PMID 15512888
- [Background] Sanchez B, Rutkove SB. Present Uses, Future Applications, and Technical Underpinnings of Electrical Impedance Myography. Curr Neurol Neurosci Rep. 2017 Sep 20;17(11):86. doi: 10.1007/s11910-017-0793-3. PMID 28933017
- [Background] Jafarpoor M, Li J, White JK, Rutkove SB. Optimizing electrode configuration for electrical impedance measurements of muscle via the finite element method. IEEE Trans Biomed Eng. 2013 May;60(5):1446-52. doi: 10.1109/TBME.2012.2237030. Epub 2013 Jan 9. PMID 23314763
- [Background] Kwon H, Malik WQ, Rutkove SB, Sanchez B. Separation of Subcutaneous Fat From Muscle in Surface Electrical Impedance Myography Measurements Using Model Component Analysis. IEEE Trans Biomed Eng. 2019 Feb;66(2):354-364. doi: 10.1109/TBME.2018.2839977. Epub 2018 May 23. PMID 29993468
- [Background] Rutkove SB. Electrical impedance myography: Background, current state, and future directions. Muscle Nerve. 2009 Dec;40(6):936-46. doi: 10.1002/mus.21362. PMID 19768754
- [Background] Rutkove SB, Aaron R, Shiffman CA. Localized bioimpedance analysis in the evaluation of neuromuscular disease. Muscle Nerve. 2002 Mar;25(3):390-7. doi: 10.1002/mus.10048. PMID 11870716
- [Background] Kowal JB, Verga SA, Pandeya SR, Cochran RJ, Sabol JC, Rutkove SB, Coates JR. Electrical Impedance Myography in Dogs With Degenerative Myelopathy. Front Vet Sci. 2022 May 27;9:874277. doi: 10.3389/fvets.2022.874277. eCollection 2022. PMID 35711791
- [Background] Wang LL, Spieker AJ, Li J, Rutkove SB. Electrical impedance myography for monitoring motor neuron loss in the SOD1 G93A amyotrophic lateral sclerosis rat. Clin Neurophysiol. 2011 Dec;122(12):2505-11. doi: 10.1016/j.clinph.2011.04.021. Epub 2011 May 25. PMID 21612980
- [Background] Li J, Yim S, Pacheck A, Sanchez B, Rutkove SB. Electrical Impedance Myography to Detect the Effects of Electrical Muscle Stimulation in Wild Type and Mdx Mice. PLoS One. 2016 Mar 17;11(3):e0151415. doi: 10.1371/journal.pone.0151415. eCollection 2016. PMID 26986564
- [Background] Pacheck A, Mijailovic A, Yim S, Li J, Green JR, McIlduff CE, Rutkove SB. Tongue electrical impedance in amyotrophic lateral sclerosis modeled using the finite element method. Clin Neurophysiol. 2016 Mar;127(3):1886-90. doi: 10.1016/j.clinph.2015.11.046. Epub 2015 Dec 11. PMID 26750579
- [Background] Shellikeri S, Yunusova Y, Green JR, Pattee GL, Berry JD, Rutkove SB, Zinman L. Electrical impedance myography in the evaluation of the tongue musculature in amyotrophic lateral sclerosis. Muscle Nerve. 2015 Oct;52(4):584-91. doi: 10.1002/mus.24565. Epub 2015 Jun 3. PMID 25580728
- [Background] Mcilduff CE, Yim SJ, Pacheck AK, Rutkove SB. Optimizing electrical impedance myography of the tongue in amyotrophic lateral sclerosis. Muscle Nerve. 2017 Apr;55(4):539-543. doi: 10.1002/mus.25375. Epub 2016 Dec 26. PMID 27511962
- [Background] Rutkove SB, Caress JB, Cartwright MS, Burns TM, Warder J, David WS, Goyal N, Maragakis NJ, Clawson L, Benatar M, Usher S, Sharma KR, Gautam S, Narayanaswami P, Raynor EM, Watson ML, Shefner JM. Electrical impedance myography as a biomarker to assess ALS progression. Amyotroph Lateral Scler. 2012 Sep;13(5):439-45. doi: 10.3109/17482968.2012.688837. Epub 2012 Jun 7. PMID 22670883
- [Background] Li J, Sung M, Rutkove SB. Electrophysiologic biomarkers for assessing disease progression and the effect of riluzole in SOD1 G93A ALS mice. PLoS One. 2013 Jun 6;8(6):e65976. doi: 10.1371/journal.pone.0065976. Print 2013. PMID 23762454
- [Background] Shefner JM, Rutkove SB, Caress JB, Benatar M, David WS, Cartwright MS, Macklin EA, Bohorquez JL. Reducing sample size requirements for future ALS clinical trials with a dedicated electrical impedance myography system. Amyotroph Lateral Scler Frontotemporal Degener. 2018 Nov;19(7-8):555-561. doi: 10.1080/21678421.2018.1510008. Epub 2018 Sep 28. PMID 30265154
- [Background] Rutkove SB, Narayanaswami P, Berisha V, Liss J, Hahn S, Shelton K, Qi K, Pandeya S, Shefner JM. Improved ALS clinical trials through frequent at-home self-assessment: a proof of concept study. Ann Clin Transl Neurol. 2020 Jul;7(7):1148-1157. doi: 10.1002/acn3.51096. Epub 2020 Jun 9. PMID 32515889
- [Background] Kapur K, Nagy JA, Taylor RS, Sanchez B, Rutkove SB. Estimating Myofiber Size With Electrical Impedance Myography: a Study In Amyotrophic Lateral Sclerosis MICE. Muscle Nerve. 2018 Nov;58(5):713-717. doi: 10.1002/mus.26187. Epub 2018 Sep 2. PMID 30175407
- [Background] Pandeya SR, Nagy JA, Riveros D, Semple C, Taylor RS, Mortreux M, Sanchez B, Kapur K, Rutkove SB. Estimating myofiber cross-sectional area and connective tissue deposition with electrical impedance myography: A study in D2-mdx mice. Muscle Nerve. 2021 Jun;63(6):941-950. doi: 10.1002/mus.27240. Epub 2021 Apr 7. PMID 33759456
- [Background] Pandeya SR, Nagy JA, Riveros D, Semple C, Taylor RS, Mortreux M, Sanchez B, Kapur K, Rutkove SB. Predicting myofiber cross-sectional area and triglyceride content with electrical impedance myography: A study in db/db mice. Muscle Nerve. 2021 Jan;63(1):127-140. doi: 10.1002/mus.27095. Epub 2020 Oct 28. PMID 33063867
- [Background] Rutkove SB, Caress JB, Cartwright MS, Burns TM, Warder J, David WS, Goyal N, Maragakis NJ, Benatar M, Sharma KR, Narayanaswami P, Raynor EM, Watson ML, Shefner JM. Electrical impedance myography correlates with standard measures of ALS severity. Muscle Nerve. 2014 Mar;49(3):441-3. doi: 10.1002/mus.24128. Epub 2013 Dec 19. PMID 24273034
- [Background] Manjaly ZR, Scott KM, Abhinav K, Wijesekera L, Ganesalingam J, Goldstein LH, Janssen A, Dougherty A, Willey E, Stanton BR, Turner MR, Ampong MA, Sakel M, Orrell RW, Howard R, Shaw CE, Leigh PN, Al-Chalabi A. The sex ratio in amyotrophic lateral sclerosis: A population based study. Amyotroph Lateral Scler. 2010 Oct;11(5):439-42. doi: 10.3109/17482961003610853. PMID 20225930